CLINICAL TRIAL: NCT03343093
Title: Restore: Improving Sexual Outcomes of Gay and Bisexual Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SPH-2018-26507; 1R01CA218657-01 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Prostatic Neoplasm
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Evaluation Control Group (Experimental): Surveys at 3 month intervals
  Interventions: Behavioral: Control
- Intervention Evaluation Test Group (Experimental): We will evaluate the effects of an educational, tailored, online rehabilitation program addressing sexual and urinary outcomes after treatment by surveying at 3 month intervals
  Interventions: Behavioral: Restore Rehabilitation Program

INTERVENTIONS:
Behavioral: Restore Rehabilitation Program — Multi-component, structured, biopsychosocial, online interactive program to address the sexual and urinary effects of prostate cancer treatment
  Arms: Intervention Evaluation Test Group
Behavioral: Control — usual care, surveys every 3 months
  Arms: Intervention Evaluation Control Group

SUMMARY:
Development and evaluation of an online intervention addressing sexual functioning in gay and bisexual men (GBM) after prostate cancer treatment.

DETAILED DESCRIPTION:
This study advances research in three areas.

First, prostate cancer is the second most common cancer among gay, bisexual, and other men who have sex with men with documented disparities, yet it is severely under-researched. Because gay sex differs from vaginal sex, physiologically; the results from 614 studies focused on heterosexual men likely do not generalize to gay and bisexual men(GBM) with prostate cancer. There have been no rehabilitation studies specific to GBM survivors of prostate cancer, so clinicians have no relevant studies to inform best practice with their GBM patients.

Second, most prostate cancer studies have tested one or rehabilitation components. The investigators will conduct the first treatment study of a state of clinical practice comprehensive rehabilitation program on GBM's quality of life, including on both urinary and sexual function and bother measures.

Third, almost all prostate cancer studies have focused on men recently treated for prostate cancer.

The long-term objective of this research is to improve the health of gay and bisexual survivors of Prostate cancer and to provide an evidence base for rehabilitation. The Investigators will develop an online rehabilitation program tailored for GBM that addresses both the sexual and urinary effects of prostate cancer treatment. In addition, The Investigators will conduct a comparative recruitment study to identify best methods to recruit 450 GBM with Prostate cancer.

Finally, the Investigators will evaluate the effects of the tailored rehabilitation program on sexual and urinary outcomes. The Investigators will conduct a 24 month, randomized controlled trial of structured rehabilitation versus routine care. The Investigators will study both GBM recently treated (last 2 years) and GBM post-treatment (2+ years), using a stratified design. This randomized control trial will identify whether a structured rehabilitation program is effective in addressing the major sexual and urinary problems caused by Prostate cancer treatment. As the first treatment study to focus on GBM with Prostate cancer (and also on oral and anal sex), it addresses a long-standing health disparity.

The study has high potential to transform rehabilitation for GBM with Prostate cancer, provide a critical evidence base for clinicians, and inform rehabilitation outcomes for all Prostate cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Gay or Bisexual Men, defined as a biological adult male, who by self-report, has had sex with a man.
2. Treated for prostate cancer, defined as (i) having been diagnosed with prostate cancer and measured by being able to report a Prostate- Specific Antigen and Gleason score; and (ii) treated by radical prostatectomy, radiation or systemically.
3. Has recent problems with sexual and/or urinary function, by self-report. This is measured by a screener item(s) asking the enrollee to describe their current function (last 4 weeks) and validated by nurse interview.
4. Internet-using
5. Living in the US (including territories) as measured by valid US zip code
6. A unique, validated individual, as measured by our published de-duplication and cross-validation protocols,230-232 and confirmed by video or phone interview.

Exclusion Criteria:

1. No Nerve Sparing and Salvage therapy.
2. Medical contraindications as determined by investigators at screening
3. Heavy smoking: more than 10 cigarettes, cigars, e-cigarettes, snuff pipe or similar product on an average day (screened over last 7 days)
4. Heavy alcohol use: more than 4 drinks per day, on two or more days, last 7 days
5. Participation is limited to English speakers/readers since intervention materials and surveys are in English.
6. Cognitive impairment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male bodied persons at risk of prostate cancer
Enrollment: 403 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Simon Rosser, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Twin Cities Campus, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosser BRS, Polter EJ, Chandiramani N, Cahill S, Wheldon CW, Konety BR, Ryan CJ, Haggart R, Kapoor A. Acceptability and Feasibility of Collecting Sexual Orientation and Expanded Gender Identity Data in Urology and Oncology Clinics. LGBT Health. 2021 Aug-Sep;8(6):420-426. doi: 10.1089/lgbt.2020.0256. Epub 2021 Aug 4. PMID 34348045

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Evaluation Control Group | Intervention Evaluation Test Group
Started | 199 | 204
Completed | 180 | 175
Not Completed | 19 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Evaluation Control Group | Intervention Evaluation Test Group | Total
Number analyzed (Participants) | 197 | 204 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (6.6) | 64 (6.7) | 63.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 197 | 204 | 401
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 13 | 22
  White | 179 | 186 | 365
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Urinary Function Scores
Description: The Urinary Function domain of the Expanded Prostate Cancer Index Composite (EPIC-50) scale was used to assess the frequency of urinary symptoms. Scores range from 0 to 100, with higher scores indicating less frequency of urinary symptoms.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale (0-100)
Arm/Group | Intervention Evaluation Control Group | Intervention Evaluation Test Group
Number analyzed (Participants) | 197 | 204
Scores on a scale (0-100) | 80.1 [78.1 to 82.2] | 81.4 [79.4 to 83.5]

2. Primary Outcome: Sexual Functioning Scores
Description: The Sexual Functioning domain of the Expanded Prostate Cancer Index Composite (EPIC-50) scale was used to assess the frequency of sexual functioning symptoms. Scores range from 0 to 100, with higher scores indicating less frequency of sexual functioning symptoms.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale (0-100)
Arm/Group | Intervention Evaluation Control Group | Intervention Evaluation Test Group
Number analyzed (Participants) | 197 | 204
Scores on a scale (0-100) | 37.5 [34.7 to 40.3] | 36.7 [33.9 to 39.4]

3. Primary Outcome: Intervention Acceptability
Description: Acceptability was measured by how much intervention group participants would recommend the intervention to a friend (if he had prostate cancer). This single Likert-type item has five response options from 1=strongly agree to 5= strongly disagree. Acceptability will be measured by adding those who answered 1=strongly agree or 2=agree on this item.
Time Frame: 3-month follow-up
Population: Percent frequencies of those rating the intervention as acceptable
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Evaluation Test Group: Acceptability was measured by how much intervention group participants thought about the intervention content, would recommended the intervention to a friend, and liked the intervention being tailored to SGM as measured by 5-point Likert items. Satisfaction with the intervention content was measured by adapting EDITS.
Arm/Group | Intervention Evaluation Test Group
Number analyzed (Participants) | 183
Participants | 156

4. Primary Outcome: Intervention Feasibility
Description: Feasibility will be measured by monitoring the number of intervention participants who could access the intervention webpage at least once within the first three months of the study.
Time Frame: 3-month follow-up
Population: Percent participants who where able to access the intervention at least once.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Evaluation Test Group: Feasibility was measured as the number of intervention participants who received the study aids and accessed the intervention website.
Arm/Group | Intervention Evaluation Test Group
Number analyzed (Participants) | 204
Participants | 189

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire 24-month trial period, beginning when the first participant accessed study materials until the last participant returned the 24-month survey.
Arm/Group | Intervention Evaluation Control Group | Intervention Evaluation Test Group
All-Cause Mortality (participants affected / at risk) | 4/197 | 4/204
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/204
Other Adverse Events (participants affected / at risk) | 0/197 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03343093/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03343093/SAP_001.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03343093/ICF_002.pdf